CLINICAL TRIAL: NCT04050761
Title: A French Prospective, Non-interventional Research ( NIR) of Nivolumab in Patients With Squamous Cell Carcinoma of the Head and Neck (SCCHN) Progressing on or After a Platinum-based Therapy
Brief Title: A Study of Nivolumab in Patients With Head and Neck Cancer.
Acronym: ProNiHN
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-9T9
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Head and Neck Cancer; Head and Neck Carcinoma; Cancer of the Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monotherapy: Participants diagnosed with recurrent or metastatic squamous cell carcinoma of the Head and Neck and whose physician has decided to initiate a treatment with Nivolumab for the first time for the treatment of SCCHN.
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on Specific Days

SUMMARY:
A prospective real world evidence study of Nivolumab use in France in patient with recurrent or metastatic squamous cell carcinoma of the Head and Neck progressing on or after a platinum based therapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Squamous Cell Carcinoma Head and Neck (SCCHN) patients progressing on or after platinum-based therapy.
* Diagnosis of SCCHN has been confirmed by histology or cytology (either at initial diagnosis or any time later during the course of the disease)
* Treatment decision to initiate a treatment with nivolumab for the first time for the treatment of SCCHN (according to the label approved in France) has already been taken

Exclusion Criteria:

* Patients previously treated with Nivolumab, Ipilimumab, or any other antibody or drug specifically targeting T-Cell Co stimulation or immune Checkpoint pathway.
* Patients currently included in an interventional clinical trial for their SCCHN.

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who are at least 18 years of age with the diagnosis of Squamous Cell Carcinoma Head and Neck that the physician has already decided to initiate a treatment with nivolumab for the first time.
Sampling Method: Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 Years

SECONDARY OUTCOMES:
Overall Survival within Sub groups | 3 year
Progression-free survival (PFS) | 3 Years
Overall response rate (ORR) | 3 years
Best overall response rate (BORR) | 3 years
Time to response (TTR) | 3 years
Duration of response (DOR) | 3 years
Incidents of Adverse Events (AEs) | 3 years
Incidents of immune-related Adverse Events | 3 years
Incident of treatment-related Adverse Events | 3 years
Number of socio-demographic characteristics in adult patients with SCCHN | 3 years
Number of clinical characteristics in adult patients with SCCHN | 3 Years
Number of treatment characteristics in adult patients with SCCHN | 3 Years
Functional Assessment of Cancer Therapy - Head & Neck (FACT-H&N) Score | 3 Years
Quality of life of caregiver (CarGoQoL ) Score | 3 Years
Supportive Care Needs Survey for Partners and Caregivers (SCNS-P&C) Assessment score | 3 Years
European Quality of Life-5 Dimensions (EQ-5D) score | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Paris, Île-de-France Region, France

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html